CLINICAL TRIAL: NCT00844571
Title: The Effectiveness of an E-learning Program About Child Maltreatment for Nurses on an A&E Department: a Randomised Controlled Trial
Brief Title: Effect E-learning Program About Child Maltreatment
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: UMC Utrecht (Other)
Collaborators: a private, non-commercial foundation that wishes to not be named (Ambiguous)
Responsible Party: Patricia Ohlsen, projectleider, Augeo-foundation
Other Study IDs: 170883
Record Dates: First submitted 2009-02-12; First posted 2009-02-16 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Child Abuse
Keywords: child abuse and neglect; child maltreatment; non accidental injury; training; educational program

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- E-learning program: Participants are committed to accomplish the program in approximately 2 hours. Additionally to these mandatory hours, they were able to access the e-learning program at any time and place.
  Interventions: Other: E-learning program
- control group

INTERVENTIONS:
Other: E-learning program — Participants are committed to accomplish the program in approximately 2 hours. Additionally to these mandatory hours, they were able to access the e-learning program at any time and place.
  Other Names: Electronic learning; Web-based learning
  Groups: E-learning program

SUMMARY:
The purpose of this study is to determine whether the e-learning program about the recognition of child maltreatment is effective in nurses on the A&E department compared to a control group.

DETAILED DESCRIPTION:
Child abuse and neglect represents an international problem with high prevalence and unacceptable levels of morbidity and mortality. Many children are seen each day in the accident and emergency departement of an hospital. Therefore the A&E departement have an important role in the identification of child maltreatment. The lack of an effective teaching program together with the failures in the child protection process has encouraged the development of a clinical-practice-oriented e-learning program on detecting child maltreatment. We will investigate the effect of this e-learning program.

ELIGIBILITY:
Inclusion Criteria:

* Working at the A&E department of the UMC-Utrecht.

Exclusion Criteria:

* Absent during one of the two measurement periods.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Nurses working at the A&E department of UMC-Utrecht
Sampling Method: Probability Sample
Enrollment: 38 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-04 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Clinical behaviour on the A&E department, self-efficacy of the nurse in the detection of child abuse and assessment of the individual performance on screening child abuse. | 2-3 months

CONTACTS AND LOCATIONS:
Overall Officials: Keetie Smeekens, Drs., Principal Investigator — UMC Utrecht

REFERENCES:
- [Derived] Walsh K, Eggins E, Hine L, Mathews B, Kenny MC, Howard S, Ayling N, Dallaston E, Pink E, Vagenas D. Child protection training for professionals to improve reporting of child abuse and neglect. Cochrane Database Syst Rev. 2022 Jul 5;7(7):CD011775. doi: 10.1002/14651858.CD011775.pub2. PMID 35788913
- [Derived] Smeekens AE, Broekhuijsen-van Henten DM, Sittig JS, Russel IM, ten Cate OT, Turner NM, van de Putte EM. Successful e-learning programme on the detection of child abuse in emergency departments: a randomised controlled trial. Arch Dis Child. 2011 Apr;96(4):330-4. doi: 10.1136/adc.2010.190801. Epub 2011 Jan 12. PMID 21233084